CLINICAL TRIAL: NCT05339230
Title: A Randomized Phase 2 and Pilot Pharmacodynamic Trial Investigating the Effect of Salovum™ and SPC-flakes on Dihydropyrimidine Induced Gastrointestinal Toxicity and Tumour Perfusion in Colorectal Cancer
Brief Title: Role of Antisecretory Factor in Dihydropyrimidine Treatment of Colorectal Cancer
Acronym: SALFLADMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: Lantmännen AB (Unknown); Sjöbergstiftelsen (Unknown); Onkologiska klinikens forskningsfond (Unknown); Swedish Cancer Society (Other)
Responsible Party: Principal Investigator, Peter Nygren, Professor in oncology, consultant in oncology, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASF 2
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Dihydropyrimidine Induced Gastrointestinal Toxicity in Colorectal Cancer
Keywords: Dihydropyrimidine; Diarrhoea; Colorectal cancer; Antisecretory factor
MeSH Terms: conditions — Diarrhea; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel 2 group randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo study products similar to the active products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Salovum egg powder high in antisecretory factor, 4 g/sachet. Four sachets, ie 16 g q 8 h for 6 days starting 6 days before 1st cycle of chemotherapy. SPC-flakes flat dose of 75 g/d divided in 2 - 4 doses started in parallel with Salovum to be continued during the first 8 weeks of chemotherapy.
  Interventions: Dietary Supplement: Salovum and SPC-flakes active or placebo
- Control (Placebo Comparator): Salovum placebo powder without antisecretory factor, 4 g/sachet. Four sachets, ie 16 g q 8 h for 6 days starting 6 days before 1st cycle of chemotherapy. SPC placebo flakes flat dose of 75 g/d divided in 2 - 4 doses started in parallel with Salovum placebo to be continued during the first 8 weeks of chemotherapy.
  Interventions: Dietary Supplement: Salovum and SPC-flakes active or placebo

INTERVENTIONS:
Dietary Supplement: Salovum and SPC-flakes active or placebo — Foods for specific medical purposes or corresponding placebo

SUMMARY:
One debilitating, and sometimes even life-threatening, toxicity from dihydropyrimidines, e g 5-FU and capecitabine, is gastrointestinal mucositis resulting in, eg severe diarrhoea necessitating in-hospital care including periods of support with iv fluids. The efficacy of current treatment for this adverse effect include iv fluids, loperamide and opioids po and octreotide sc is moderate and new treatment principles or, preferably, ways to prevent such toxicity, are urgently needed. Cholera induced diarrhoea, as well as other forms of diarrhoea-inducing agents, has been shown to elicit a stimulated, endogenous production of a protein, named "antisecretory factor", ASF. ASF acts by modulating secretion of water and ions but also counteracts inflammatory processes.

ASF is also produced by hens fed on a diet of fermented grains or a specific diet of sugars and amino acids, leading to an accumulation of the ASF protein in the egg yolk. Spray dried yolk in the form of a powder is commercialized as Salovum registered by the EU authorities as "Food for specific medical purposes". Another way to increase ASF and, thus, to achieve benefit, is to induce its production/ conversion by ingestion of oat flakes, specially processed (similar to malting) to contain the proper mix of sugars and amino acids. Such flakes are also commercially available (SPC-flakes) as "Food for specific medical purposes".

Salovum has been shown to rapidly, ie within hours to a few days, antagonize diarrhoeal diseases of various etiologies. It has also been used against high fluid passages and inflammation in Crohns disease, Colitis ulcerosa and carcinoids in adults. SPC-flakes have similar effects but need weeks of administration to emerge. Interestingly from an oncological perspective, provision of exogenous ASF and induction of endogenous ASF has been shown to reduce interstitial fluid pressure (IFP) in tumours, increase tumour uptake of cytotoxic drugs and improve survival in animal tumour models.

With this background the present study will investigate if administration of ASF in the form of Salovum combined with induction of endogenous ASF by intake of SPC-flakes might be beneficial in colorectal cancer (CRC) patients to prevent dihydropyrimidine based chemotherapy induced gastrointestinal mucositis and to reduce tumor interstitial fluid pressure .

DETAILED DESCRIPTION:
The pyrimidine analogue 5-fluorouracil (5-FU) has a history in oncology for more than 50 years, and is still the backbone in chemotherapy regimens, in particular for gastrointestinal cancer although it is now often substituted with the oral prodrug capecitabine. Since colorectal cancer is the third most common cancer in Europe and the US a great number of patients will be exposed to 5-FU either as part of a curative intent, ie (neo)adjuvant, or with a palliative intention.

One debilitating, and sometimes even life-threatening, toxicity from dihydropyrimidines, e g 5-FU and capecitabine, is gastrointestinal mucositis resulting in, eg severe diarrhoea necessitating in-hospital care including periods of support with iv fluids. The efficacy of current treatment for this adverse effect include iv fluids, loperamide and opioids po and octreotide sc is moderate and new treatment principles or, preferably, ways to prevent such toxicity, are urgently needed. Mucositis is a common adverse effect also from a number of other cancer drugs as well as from radiotherapy.

Cholera induced diarrhoea, as well as other forms of diarrhoea-inducing agents, has been shown to elicit a stimulated, endogenous production of a protein, named "antisecretory factor", ASF. This protein has been chemically characterized in detail. ASF acts by modulating secretion of water and ions but also counteracts inflammatory processes. One of the biologically active peptides of the ASF protein is AF 16, a 16 amino acids long peptide which can easily be synthesized, is chemically very stable, and is therefore used for experimental purposes.

ASF is also produced by hens fed on a diet of fermented grains or a specific diet of sugars and amino acids, leading to an accumulation of the ASF protein in the egg yolk. Spray dried yolk in the form of a powder is commercialized as Salovum registered by the EU authorities as "Food for specific medical purposes", i e is not a drug from a regulatory perspective. Therefore, clinical studies with Salovum (or SPC-flakes, see below) do not need approval from the Medical Products Agency.

Salovum rapidly increase the plasma ASF-concentration. Another way to increase ASF and, thus, to achieve benefit, is to induce its production/conversion by ingestion of oat flakes, specially processed (similar to malting) to contain the proper mix of sugars and amino acids. Such flakes are also commercially available (SPC-flakes) as "Food for specific medical purposes" and has been recommended or considered for a number of secretory pathological conditions, e g for treatment of Mb Meniére.

Salovum has been shown to rapidly, ie within hours to a few days, antagonize diarrhoeal diseases of various etiologies. It has also been used against high fluid passages and inflammation in Crohns disease, Colitis ulcerosa and carcinoids in adults. SPC-flakes have similar effects but need weeks of administration to emerge. Importantly, to raise body ASF, by Salovum or SPC-flakes, for the above indications has not been associated with adverse effects.

Interestingly from an oncological perspective, provision of exogenous ASF and induction of endogenous ASF has been shown to reduce interstitial fluid pressure (IFP) in tumours, increase tumour uptake of cytotoxic drugs and improve survival in animal tumour models.

Thus, to raise body ASF by administration of ASF in the form of Salovum or its endogenous induction by SPC-flakes is seemingly a promising strategy worthwhile to investigate in cancer, both for treatment and counteraction of adverse effects, notably gastrointestinal mucositis, and for improvement of drug cancer treatment. While a clinical trial on administration of ASF as a strategy to improve cancer therapy, notably in glioblastoma, is in a pilot early phase, there is no study ongoing with the aim to counteract chemotherapy induced mucositis.

With this background the present study will investigate if administration of ASF in the form of Salovum combined with induction of endogenous AF by intake of SPC-flakes might be beneficial in colorectal cancer (CRC) patients to prevent dihydropyrimidine based chemotherapy induced gastrointestinal mucositis. Since the study team has also experience from measurements in patients of tumour IFP using 15O-labeled water PET, a pharmacodynamic pilot study for assessement of Salovum/SPC induced changes in tumour IFP will be included as an add on to the main study and open for 10 patients with liver metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically confirmed diagnosis of colorectal cancer.
3. Planned to start 1st line dihydropyrimidine (i e 5-FU or capecitabine) based chemotherapy in the adjuvant, neoadjuvant or palliative setting.
4. Planned duration of chemotherapy ≥ 2 months.
5. Signed informed consent.
6. Liver metastatic disease (pharmacodynamics study only).

Exclusion Criteria:

1. Contraindications to the investigational product, e g known or suspected hypersensitivity to the investigational products or expected inability to their use in accordance with the protocol.
2. Lack of suitability for participation in the study, e g expected difficulties to follow the protocol procedures, as judged by the investigator.
3. Prior exposure to 5-FU based chemotherapy.
4. Prior exposure to Salovum or SPC-flakes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of diarrhoea CTCAEv5.0 ≥ grade 2. | During first 2 months of chemotherapy
  Chemotherapy induced toxicity to be counteracted by intervention

SECONDARY OUTCOMES:
Incidence of in-patient care for chemotherapy induced gastrointestinal mucositis including number of days in hospital and with parenteral fluids. | During first 2 months of chemotherapy
  Chemotherapy induced toxicity to be counteracted by intervention
Change from baseline in patient reported hQoL and abdominal symptoms assessed by EORTC QLQ-30 and the colorectal cancer specific Q29 subscale. | During first 2 months of chemotherapy
  Patient reported chemotherapy induced toxicity to be counteracted by intervention
Incidence and severity of other chemotherapy induced adverse effects according to CTCAEv5.0. | During first 2 months of chemotherapy
  Chemotherapy induced toxicity to be counteracted by intervention
Increase in P-ASF concentration from baseline to day 7 from start of investigational product/placebo and just prior to treatment cycle 2, 3 and 4 (as applicable). | During first 2 months of chemotherapy
  To reflect study products pharmacodynamics and patient compliance
Relationships between P-ASF concentration and adverse effects. | During first 2 months of chemotherapy
  Assessment of biomarker related to potential benefit
Tumour response rate according to RECIST v1.1 (locally advanced and metastatic settings only). | At 1st radiological tumor response evaluation, approximately 2 months from start of chemotherapy
  Assessment of benefit, if any, from ASF elevation on drug efficacy
Incidence of adverse events CTCAEv5.0 grade ≥ 3 considered probably related to investigational products/placebo. | During first 2 months of chemotherapy
  Assessment of study product safety when combined with chemotherapy

OTHER OUTCOMES:
Change in liver metastasis water perfusion. | One week prior to start of chemotherapy
  Assessment of change in tumor interstitial fluid pressure by antisecretory factor
Change in liver metastasis tumor blood flow. | One week prior to start of chemotherapy
  Assessment of change in tumor interstitial fluid pressure by antisecretory factor

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
To be considered.

REFERENCES:
- [Background] Ulgheri C, Paganini B, Rossi F. Antisecretory factor as a potential health-promoting molecule in man and animals. Nutr Res Rev. 2010 Dec;23(2):300-13. doi: 10.1017/S0954422410000193. Epub 2010 Aug 5. PMID 20684797
- [Background] Johansson E, Jennische E, Lange S, Lonnroth I. Antisecretory factor suppresses intestinal inflammation and hypersecretion. Gut. 1997 Nov;41(5):642-5. doi: 10.1136/gut.41.5.642. PMID 9414971
- [Background] Zaman S, Aamir K, Lange S, Jennische E, Silfverdal SA, Hanson LA. Antisecretory factor effectively and safely stops childhood diarrhoea: a placebo-controlled, randomised study. Acta Paediatr. 2014 Jun;103(6):659-64. doi: 10.1111/apa.12581. Epub 2014 Mar 10. PMID 24484450
- [Background] Bjorck S, Bosaeus I, Ek E, Jennische E, Lonnroth I, Johansson E, Lange S. Food induced stimulation of the antisecretory factor can improve symptoms in human inflammatory bowel disease: a study of a concept. Gut. 2000 Jun;46(6):824-9. doi: 10.1136/gut.46.6.824. PMID 10807895
- [Background] Al-Olama M, Wallgren A, Andersson B, Gatzinsky K, Hultborn R, Karlsson-Parra A, Lange S, Hansson HA, Jennische E. The peptide AF-16 decreases high interstitial fluid pressure in solid tumors. Acta Oncol. 2011 Oct;50(7):1098-104. doi: 10.3109/0284186X.2011.562240. Epub 2011 Mar 4. PMID 21375367
- [Background] Ilkhanizadeh S, Sabelstrom H, Miroshnikova YA, Frantz A, Zhu W, Idilli A, Lakins JN, Schmidt C, Quigley DA, Fenster T, Yuan E, Trzeciak JR, Saxena S, Lindberg OR, Mouw JK, Burdick JA, Magnitsky S, Berger MS, Phillips JJ, Arosio D, Sun D, Weaver VM, Weiss WA, Persson AI. Antisecretory Factor-Mediated Inhibition of Cell Volume Dynamics Produces Antitumor Activity in Glioblastoma. Mol Cancer Res. 2018 May;16(5):777-790. doi: 10.1158/1541-7786.MCR-17-0413. Epub 2018 Feb 5. PMID 29431617